CLINICAL TRIAL: NCT05900986
Title: An Open-label, Single-arm, Phase 1b/2 Study to Investigate the Safety, Efficacy and Pharmacokinetics of LS301-IT in Female Patients Undergoing Partial Mastectomy and Sentinel Lymph Node Biopsy (SLNB) for Ductal Carcinoma in Situ (DCIS) or Stage I-II Primary Invasive Breast Cancer
Brief Title: LS301-IT in Partial Mastectomy and Sentinel Lymph Node Biopsy (SLNB) for DCIS or Stage I-II Primary Invasive Breast Cancer
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Integro Theranostics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LS301-IT-B101
Record Dates: First submitted 2023-05-10; First posted 2023-06-13 (Actual); Last update posted 2025-10-16 (Actual); Status verified 2025-10

CONDITIONS: Breast Cancer; DCIS; Invasive Duct Carcinoma of Breast
MeSH Terms: conditions — Breast Neoplasms; Carcinoma, Intraductal, Noninfiltrating; Carcinoma, Ductal, Breast

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- LS301-IT (Experimental): LS301-IT will be administered by IV injection
  Interventions: Drug: LS301-IT 0.025 mg/kg; Drug: LS301-IT 0.05 mg/kg; Drug: LS301-IT 0.075 mg/kg; Drug: LS301-IT 0.1 mg/kg

INTERVENTIONS:
Drug: LS301-IT 0.025 mg/kg — The dose of LS301-IT planned to be administered to the first cohort of patients is 0.025 mg/kg. Depending on the results the dose for subsequent cohorts will be increased to 0.05, 0.075, and 0.1 mg/kg; the dose may also be decreased (by 50% as necessary). The optimal dose determined in Periods 1 and 2 will be administered to patients in Period 3.
Drug: LS301-IT 0.05 mg/kg — Depending on the results the dose for subsequent cohorts will be increased to 0.05, 0.075, and 0.1 mg/kg; the dose may also be decreased. The optimal dose determined in Periods 1 and 2 will be administered to patients in Period 3.
Drug: LS301-IT 0.075 mg/kg — Depending on the results the dose for subsequent cohorts will be increased to 0.05, 0.075, and 0.1 mg/kg; the dose may also be decreased. The optimal dose determined in Periods 1 and 2 will be administered to patients in Period 3.
Drug: LS301-IT 0.1 mg/kg — Depending on the results the dose for subsequent cohorts will be increased to 0.05, 0.075, and 0.1 mg/kg; the dose may also be decreased. The optimal dose determined in Periods 1 and 2 will be administered to patients in Period 3.

SUMMARY:
The aim of this Phase 1b/2 study is to investigate the safety, efficacy, and pharmacokinetics (PK) of a single dose of LS301-IT, a novel fluorescence imaging agent developed by Integro Theranostics (IT), administered by intravenous (IV) injection in female patients undergoing partial mastectomy for DCIS (whether or not undergoing planned SLNB) or Stage I-II primary invasive breast cancer undergoing SLNB. Safety is the primary objective of this study, followed by efficacy that will be assessed from fluorescence imaging observations and data.

DETAILED DESCRIPTION:
This is a Phase 1b/Phase 2, open-label study to investigate the use of LS301-IT (investigational medicinal product [IMP]), a fluorescence imaging agent used for visualization of tumor margins and SLNs in female patients with DCIS or Stage I-II, primary invasive carcinoma of the breast, for which the patient's primary surgical treatment is partial mastectomy.

Eligible patients will be enrolled into either:

* Phase 1b (Period 1): dose finding (escalation/de-escalation), and dose timing adjustment;
* Phase 2a (Period 2): expanded sample size based on acceptable dosing regimen, that being the dose level(s) and time interval between LS301-IT injection and surgery, determined in Period 1; or
* Period 2b (Period 3): allow surgeon to make additional surgical decisions based on fluorescence imaging findings during surgery (Period 3 will not be opened until results are available from Periods 1 and 2 and further FDA consultation is obtained).

ELIGIBILITY:
Inclusion Criteria:

* DCIS (whether or not undergoing planned SLNB) or patients with Stage I-II, primary invasive carcinoma of the breast undergoing SLNB for which the patient's primary surgical treatment is single breast partial mastectomy.
* ECOG performance status of 0 to 2

Exclusion Criteria:

* Contraindications for surgery.
* Simultaneous bilateral lumpectomies and bilateral partial mastectomies.
* History of drug-related anaphylactic reactions, including those attributed to indocyanine green (ICG) or other agents used in the study
* Prior chemotherapy, endocrine therapy, or biologic therapy for current clinically or biopsy proven breast cancer for Period 1.
* Open surgery in the ipsilateral breast within a period of 1 year before administration of LS301-IT.
* History of radiation therapy to the chest.
* The lymphatic imaging agent ICG cannot be used prior to the partial mastectomy and SLNB procedures on the day of surgery.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — female with breast cancer
Enrollment: 100 (Estimated)
Dates: Start 2023-07-14 (Actual); Primary Completion 2025-10-06 (Actual); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Adverse Events | 30 days
  Number of participants with treatment-related adverse events
Pharmacodynamics | during surgery
  Tumor to non-tumor ratio fluorescence response
Pharmacodynamics | During surgery
  Surgeon's assessment using a semi-quantitative scoring system of fluorescence compared with intraoperative and postoperative pathology assessments.
Cmax | 24 hours
  maximum observed plasma concentration main metabolite in plasma.
AUCinf | 24 hours
  area under the plasma concentration time curve from time 0 extrapolated to infinite time
AUClast | 24 hours
  area under the plasma concentration-time curve from time 0 to the last quantifiable plasma concentration
Tmax | 24 hours
  time to reach maximal plasma concentration (Tmax)
t1/2 | 24 hours
  elimination/apparent terminal elimination half life

CONTACTS AND LOCATIONS:
Overall Officials: Dan Thompson, Study Director — Integro Theranostics
Locations (9):
- United States (9):
  - Integro Theranostics Research Site #2, Scottsdale, Arizona
  - Integro Theranostics Research Site #12, Washington D.C., District of Columbia
  - Integro Theranostics Research Site #9, Weston, Florida
  - Integro Theranostics Research Site #6, The Bronx, New York
  - Integro Theranostics Clinical Research Site #8, Winston-Salem, North Carolina
  - Integro Theranostics Research Site #10, Cleveland, Ohio
  - Integro Theranostics Research Site #5, Philadelphia, Pennsylvania
  - Integro Theranostics Research Site #3, Dallas, Texas
  - Integro Theronostics Research Site #1, Houston, Texas

IPD SHARING:
Plan to Share IPD: No